CLINICAL TRIAL: NCT04106440
Title: Pilot Study of Connected Diabetes Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1447976
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Use of applications to share data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application Use (Experimental): Participants will be asked to use applications to track food intake, carbohydrate counts, insulin delivered, and blood sugar values and share the data with the study team.
  Interventions: Behavioral: Application Use
- Standard of Care (No Intervention): The control group will receive usual care during their hospitalizations at the time of diabetes diagnosis, and during the time between hospital discharge and first visit to the UCD Pediatric Diabetes clinic.

INTERVENTIONS:
Behavioral: Application Use — Use applications after initial diagnosis to share information with study team.
  Arms: Application Use

SUMMARY:
To test the hypothesis that remote sharing of health data - including measured blood glucose values as well as patient-reported carbohydrate counts and insulin doses - with the UC Davis Pediatric Diabetes team via connected health applications is feasible for pediatric patients with newly diagnosed type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with T1D in the past 6 weeks
* Daily access to the internet via a wireless connection

Exclusion Criteria:

* Does not plan to attend the UC Davis Pediatric Endocrinology clinic for future diabetes care
* Primary caregiver does not speak English

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Connected Health Survey | 1 month after diabetes diagnosis
  Parent reported survey to determine how often families review blood sugar numbers and the ease of use of the applications.
Connected Health Survey | 6 months after diabetes diagnosis
  Parent reported survey to determine how often families review blood sugar numbers and the ease of use of the applications.

SECONDARY OUTCOMES:
Frequency of blood glucose monitoring | At each clinic visit until 6 months since diagnosis
  How often patients are monitoring their blood sugar (documented in electronic medical record)
Hemoglobin A1c values | At each clinic visit until 6 months since diagnosis
  Hemoglobin A1c values collected at each clinic visit (documented in electronic medical record)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crossen S, Romero C, Reggiardo A, Michel J, Glaser N. Feasibility and Impact of Remote Glucose Monitoring Among Patients With Newly Diagnosed Type 1 Diabetes: Single-Center Pilot Study. JMIR Diabetes. 2022 Jan 17;7(1):e33639. doi: 10.2196/33639. PMID 35037887